CLINICAL TRIAL: NCT02277132
Title: The Dutch STRIDER (Sildenafil TheRapy In Dismal Prognosis Early-onset Fetal Growth Restriction)
Acronym: STRIDER
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Results of interim analysis
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other)
Responsible Party: Principal Investigator, Wessel Ganzevoort, J.W. Ganzevoort MD PhD, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 80-83600-98-20081
Record Dates: First submitted 2014-09-29; First posted 2014-10-28 (Estimated); Last update posted 2018-07-26 (Actual); Status verified 2018-07

CONDITIONS: Fetal Growth Restriction
Keywords: Fetal growth restriction; Sildenafil
MeSH Terms: conditions — Fetal Growth Retardation | interventions — Sildenafil Citrate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sildenafil (Active Comparator): Sildenafil 25 mg tablets three times daily orally from randomization until delivery
  Interventions: Drug: Sildenafil
- Placebo (Placebo Comparator): Placebo tablets three times daily orally from randomization until delivery
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Sildenafil — Sildenafil 25 mg three times daily orally from randomization until delivery
  Other Names: Viagra
  Arms: Sildenafil
Drug: Placebo — Placebo tablets three times daily orally from randomization until delivery
  Arms: Placebo

SUMMARY:
Rationale: Severe, early-onset fetal growth restriction (FGR) due to placental insufficiency is associated with a high risk of perinatal morbidity with long-lasting sequelae and mortality. Placental insufficiency is the result of abnormal formation and function of the placenta (placentation) with inadequate remodelling of the maternal spiral (uteroplacental) arteries. There is currently no therapy available with demonstrated effectiveness. Evidence suggests Sildenafil citrate improves uteroplacental blood flow, growth, and meaningful outcomes.

Objective: To evaluate the effectiveness of sildenafil (versus placebo) in achieving healthy perinatal survival.

Study design: Multicenter nationwide randomized placebo-controlled clinical trial.

Study population: Women with a singleton pregnancy between 20 and 30 weeks with severe fetal growth restriction of likely placental origin, and with estimated significant likelihood of perinatal death.

Intervention: Sildenafil 25mg or placebo tablet orally three times daily. Main study parameters/endpoints: Perinatal healthy survival, i.e. survival without severe neonatal morbidity at term age.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: Taking tablets three times daily. No additional ultrasounds, other than standard clinical protocol, one extra blood sample at inclusion. No risks anticipated, unexpected medication-associated risks can't be excluded on beforehand.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria ((I OR II) AND III):

* At 20+0-27+6 weeks: an ultrasound measurement of the fetal abdominal circumference (AC) <3rd percentile for gestational age or an ultrasound estimate of fetal weight (EFW) <5th percentile OR
* At 28+0-29+6 weeks: an ultrasound estimate of fetal weight (EFW) <700 grams using Hadlock C formula AND
* Likely placental origin defined by (a AND/OR b AND/OR c AND/OR d)

  * The presence of uterine artery notching
  * Abnormal flow velocity patterns of the umbilical artery or middle cerebral artery
  * Maternal hypertensive disorders
  * Low PlGF in point-of-care assessment

Exclusion Criteria:

* Plan to terminate pregnancy for maternal or fetal indication within days
* Known multiple pregnancy
* Identified congenital anomalies or congenital infection
* Maternal age at eligibility <18 years
* Cocaine use
* Current use of sildenafil
* Current use of cyp3A5 inhibitors: amiodaron, azitromycine, ciclosporine, claritromycine, diltiazem, erytromycine, fluconazol, itraconazol, ketoconazol, verapamil, voriconazol.
* Recent myocardial infarction or stroke

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 216 (Actual)
Dates: Start 2015-01; Primary Completion 2018-07-19 (Actual); Study Completion 2018-07-19 (Actual)

PRIMARY OUTCOMES:
Intact neonatal survival until term age | Term age, up to 20 weeks after randomization

SECONDARY OUTCOMES:
Fetal growth velocity assessed by ultrasound: abdominal circumference measurements (AC) | At contact moments with the patient, up to 20 weeks after randomization
  Average daily increase in ultrasound-estimated AC
Age-adequate performance on the two-year Bayley scales of infant development (BSID)-III (composite cognitive score and composite motor score) | 2 years corrected age, up to 2 years and three months after randomization
Co-incidence and severity of the maternal syndrome of pre-eclampsia / HELLP-syndrome (Hemolysis Elevated Liver enzymes Low Platelets) | At contact moments with the patient, up to 20 weeks after randomization

OTHER OUTCOMES:
Fetal ultrasound and Doppler studies: estimated fetal weight, abdominal circumference and Doppler of umbilical artery | At contact moments with the patients, up to 20 weeks after randomization
  Umbilical artery, middle cerebral artery, ductus venosus and aortic isthmus Doppler indices; fetal biometry; amniotic fluid index; deepest vertical amniotic fluid pocket.
PlGF (Placental Growth Factor) point-of-care assessment | At baseline
  If possible in designated clinic

CONTACTS AND LOCATIONS:
Overall Officials: J.W. Ganzevoort, MD PhD, Principal Investigator — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA); K Bloemenkamp, MD PhD, Study Chair — Leiden University Medical Center; P von Dadelszen, Prof, Study Chair — University of British Columbia; C de Groot, Prof, Study Chair — VU Medisch Centrum; M.W. de Laat, MD PhD, Study Chair — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA); B.W. Mol, Prof, Study Chair — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA); M. Porath, MD PhD, Study Chair — Perinataal Centrum MMC Veldhoven; J.A.M. van der Post, Prof, Study Chair — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA); A. van Wassenaer, MD PhD, Study Chair — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Locations (10):
- Netherlands (10):
  - Radboud Medisch Centrum Nijmegen, Nijmegen, Gelderland
  - Maastricht Universitair Medisch Centrum, Maastricht, Limburg
  - Maxima Medisch Centrum, Veldhoven, North Brabant
  - Vrije Universiteit Medisch Centrum, Amsterdam, North Holland
  - Academisch Medisch Centrum, Amsterdam, North Holland
  - Isala Klinieken, Zwolle, Overijssel
  - Leids Universitair Medisch Centrum, Leiden, South Holland
  - Erasmus Medisch Centrum Rotterdam, Rotterdam, South Holland
  - Universitair Medisch Centrum Groningen, Groningen
  - Universitair Medisch Centrum Utrecht, Utrecht

REFERENCES:
- [Derived] Pels A, Derks J, Elvan-Taspinar A, van Drongelen J, de Boer M, Duvekot H, van Laar J, van Eyck J, Al-Nasiry S, Sueters M, Post M, Onland W, van Wassenaer-Leemhuis A, Naaktgeboren C, Jakobsen JC, Gluud C, Duijnhoven RG, Lely T, Gordijn S, Ganzevoort W; Dutch STRIDER Trial Group. Maternal Sildenafil vs Placebo in Pregnant Women With Severe Early-Onset Fetal Growth Restriction: A Randomized Clinical Trial. JAMA Netw Open. 2020 Jun 1;3(6):e205323. doi: 10.1001/jamanetworkopen.2020.5323. PMID 32585017
- [Derived] Pels A, Jakobsen JC, Ganzevoort W, Naaktgeboren CA, Onland W, van Wassenaer-Leemhuis AG, Gluud C. Detailed statistical analysis plan for the Dutch STRIDER (Sildenafil TheRapy In Dismal prognosis Early-onset fetal growth Restriction) randomised clinical trial on sildenafil versus placebo for pregnant women with severe early onset fetal growth restriction. Trials. 2019 Jan 11;20(1):42. doi: 10.1186/s13063-018-3136-z. PMID 30635020
- [Derived] Pels A, Kenny LC, Alfirevic Z, Baker PN, von Dadelszen P, Gluud C, Kariya CT, Mol BW, Papageorghiou AT, van Wassenaer-Leemhuis AG, Ganzevoort W, Groom KM; international STRIDER Consortium. STRIDER (Sildenafil TheRapy in dismal prognosis early onset fetal growth restriction): an international consortium of randomised placebo-controlled trials. BMC Pregnancy Childbirth. 2017 Dec 28;17(1):440. doi: 10.1186/s12884-017-1594-z. PMID 29282009